CLINICAL TRIAL: NCT01105494
Title: Prospective Study Evaluating the Quality of Life in Dialysis Patients With End Stage Renal Disease
Brief Title: An Observational Study of Epoetin Beta [Neorecormon] to Evaluate the Quality of Life in Patients on Dialysis With Chronic Renal Anemia
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML21906
Record Dates: First submitted 2010-04-14; First posted 2010-04-16 (Estimated); Last update posted 2012-09-13 (Estimated); Status verified 2011-06

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — epoetin beta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Drug: epoetin beta [NeoRecormon] — As prescribed by physician

SUMMARY:
This multicenter, prospective, observational study will evaluate the quality of life and the factors that influence the quality of life of epoetin beta [Neorecormon] in patients with renal chronic anemia, who are on dialysis. For each eligible patient data will be collected for 6 months. Target sample size is 5000-7000 patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >/=18 years of age
* Dialysis patients with chronic renal anemia
* Written informed consent

Exclusion Criteria:

* Red blood cell transfusion in the previous 2 months
* Severe neuropsychological disorder
* Diabetic patients with serious complications

This trial is being conducted in Morocco.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dialysis patients with end-stage kidney disease on treatment with epoetin beta [Neorecormon]
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Actual)
Dates: Start 2008-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Quality of life assessment: Kidney Disease Quality of Life Questionnaire | Throughout study: 6 months

SECONDARY OUTCOMES:
Evaluation of factors (demographic and social characteristics, dialysis method) influencing the quality of life | Throughout study: 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Casablanca, Morocco